CLINICAL TRIAL: NCT03160521
Title: Multicenter, Randomized, Double-Blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Intramuscular Injections of Risperidone ISM® in Patients With Acute Exacerbation of Schizophrenia
Brief Title: Study to Evaluate the Efficacy and Safety of Risperidone in Situ Microparticle (ISM)® in Patients With Acute Schizophrenia
Acronym: PRISMA-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rovi Pharmaceuticals Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ROV-RISP-2016-01
Record Dates: First submitted 2017-05-12; First posted 2017-05-19 (Actual); Results first posted 2022-02-04 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-01

CONDITIONS: Acute Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study drug will be administered under double-blind conditions so that investigators, site staff, and patients will not be aware about the identity of the study drug (ie, blinded Risperidone ISM 75 mg, Risperidone ISM 100 mg, or placebo) administered to any given patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Risperidone ISM 75 mg (Experimental): Patients assigned to this arm will received 75 mg of Risperidone ISM during double-blind treatment period.
  Interventions: Drug: Risperidone ISM 75 mg
- Risperidone ISM 100 mg (Experimental): Patients assigned to this arm will received 100 mg of Risperidone ISM during double-blind treatment period.
  Interventions: Drug: Risperidone ISM 100 mg
- Placebo (Placebo Comparator): Patients assigned to this arm will received placebo of Risperidone ISM during double-blind treatment period.
  Interventions: Drug: Placebo of Risperidone ISM

INTERVENTIONS:
Drug: Risperidone ISM 75 mg — Monthly (once every 4 weeks) IM injection in the gluteal or deltoid muscle.
  Other Names: Risperidone ISM
  Arms: Risperidone ISM 75 mg
Drug: Risperidone ISM 100 mg — Monthly (once every 4 weeks) IM injection in the gluteal or deltoid muscle.
  Other Names: Risperidone ISM
  Arms: Risperidone ISM 100 mg
Drug: Placebo of Risperidone ISM — Monthly (once every 4 weeks) IM injection in the gluteal or deltoid muscle.
  Other Names: PLACEBO
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study designed to evaluate the efficacy and safety of intramuscular (IM) injections of Risperidone ISM® (75 or 100 mg) or placebo, in patients with acute exacerbation of schizophrenia.

DETAILED DESCRIPTION:
The study design includes a screening period, a 12-week treatment period, and a follow-up period. Eligible patients will be randomly assigned, under double-blind conditions, to receive the following study drug treatments in a 1:1:1 ratio during the double-blind treatment period: Risperidone ISM® 75 mg, Risperidone ISM® 100 mg, or placebo. The IM study drug (double-blind active Risperidone ISM® or placebo) will be administered in a deltoid or gluteal muscle for a total of 3 times, once every 4 weeks, during the 12-week treatment period.

If indicated for an individual patient, prohibited medications may be washed out during the screening period. Patients who have never taken Risperidone must have a brief trial of oral Risperidone in order to ensure a lack of any clinically significant hypersensitivity reactions before the first dose of the study drug is administered.

Efficacy will be assessed by describing changes in scores on standard psychiatric assessment tools at each visit. Safety assessments will also be conducted at each visit.

The primary objective of this study is the following:

• To evaluate the efficacy of Risperidone ISM as compared with that of placebo in the treatment of patients with acute exacerbation of schizophrenia

The secondary objectives of this study are the following:

* To characterize safety and tolerability of Risperidone ISM as compared with that of placebo in patients with acute exacerbation of schizophrenia
* To quantify healthcare resource utilization (HRU), health-related quality of life (HRQL), and social functioning in patients treated with Risperidone ISM versus placebo for an acute exacerbation of schizophrenia
* To explore pharmacokinetic characteristics of Risperidone ISM and associations with efficacy

Patients who complete planned double-blind study drug treatments and study evaluations may be eligible to participate in an optional long-term extension segment of the study in which treatment with open-label Risperidone ISM 75 or 100 mg (randomly assigned) would begin immediately; for patients who do not participate in the extension segment, a safety follow-up phone contact will occur after the end-of-treatment visit.

In addition to patients continuing from the double-blind segment of the study (rollover patients), patients not previously enrolled in the study (de novo patients) may be eligible to enter the long-term extension segment of the study. These patients will be evaluated for eligibility at a screening visit and, if eligible, will be allocated to receive either 75 or 100 mg Risperidone ISM every 4 weeks for approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for enrolment into the study, each patient must meet all of the following criteria at screening:

1. Capable of providing informed consent

   1. A signed informed consent form must be provided before any study assessments are performed
   2. Patients must be fluent in the language that is spoken by the investigator and the study site staff (including raters) and must be able to read and understand the words in which the informed consent is written
2. Age ≥ 18 and ≤ 65 years
3. Body mass index 18.5 to 40.0 kg/m2 (inclusive)
4. Current diagnosis of schizophrenia, according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria

   1. Currently experiencing an acute exacerbation or relapse with onset < 2 months before screening
   2. If inpatient at screening, has been hospitalized for < 2 weeks for the current exacerbation
   3. ≥ 2 years have elapsed since initial onset of active-phase schizophrenia symptoms
5. Has been able to achieve outpatient status for > 4 months during the past year
6. Has previously had a clinically significant beneficial response (improvement in schizophrenia symptoms), as determined by the investigator, to treatment with an antipsychotic medication other than clozapine
7. Agrees to discontinue prohibited medications as applicable and as clinically indicated according to investigator instructions
8. Dosages of all permitted medications are considered to have been stable (with the exception of medication to be used on an as-needed basis) for ≥ 2 weeks prior to the baseline visit and to remain stable during participation in this study
9. Positive and Negative Syndrome Scale (PANSS) results at the screening and baseline visits meets the following criteria:

   a. Total score between 80 and 120, inclusive b. Score of ≥ 4 (moderate or greater) for ≥ 2 of the following Positive Scale items: i. Item 1 (P1: delusions) ii. Item 2 (P2: conceptual disorganization) iii. Item 3 (P3: hallucinatory behavior) iv. Item 6 (P6: suspiciousness/persecution)
10. Clinical Global Impression - Severity (CGI-S) score of ≥ 4 (moderately ill or worse)
11. Resides in a stable living situation and is anticipated to return to that same stable living situation after discharge from the inpatient study unit, in the opinion of the investigator
12. Has an identified reliable informant who is anticipated to remain the same after the patient is discharged from the inpatient study unit, in the opinion of the investigator
13. Meets the following criteria:

    a. If a sexually active, is using a medically accepted contraceptive method, and will continue to use such throughout participation in this study (and for ≥ 6 months after the last dose of IM study drug has been administered); acceptable methods include the following: i. Condoms (male or female) with or without a spermicidal agent ii. Diaphragm or cervical cap with spermicide iii. Intrauterine device iv. Hormonal contraceptive b. If not currently sexually active, them meets the following criteria: i. Agrees that if sexually activity resumes while participating in this study, a medically accepted contraception method will be used
14. Willing and able to be confined to an inpatient study unit for up to 2 weeks (or longer if clinically indicated), as applicable and as clinically indicated according to investigator instructions
15. Agrees not to post any personal medical data related to the study or information related to the study on any website or social media site (eg, Facebook, Twitter, and others) during the study duration

Exclusion Criteria:

An individual who meets any of the following criteria at screening will not be permitted to enroll in the study:

1. History of proven inadequate clinical response to treatment with therapeutic doses (with good compliance) of risperidone or paliperidone
2. History of treatment resistance, defined as failure to respond to 2 discrete adequate trials (≥ 4 weeks with an adequate dose) of 2 different antipsychotic medications; history of clozapine use (exception: use was not because of treatment resistance or refractory psychotic symptoms)
3. Improvement in PANSS total score 20% or greater between the initial screening visit and first injection
4. Known or suspected intolerance of or allergy or hypersensitivity to risperidone, paliperidone, or any of the excipients in the IM formulations of these
5. History of neuroleptic malignant syndrome, clinically significant tardive dyskinesia, or tardive dystonia
6. History of any other medical condition that is considered to pose any unjustifiable risk or interfere with study assessments
7. Clinically significant extrapyramidal symptoms at screening or baseline
8. Answer of "yes" on item 4 or on item 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) (ideation) with the most recent episode occurring within the past 2 months, or answer "yes" to any of the 5 items (behavior) with an episode occurring within the last year
9. Current diagnosis or a history of substance use disorder according to DSM-5 criteria within 6 months prior to the screening visit (with the exception of tobacco, mild cannabis, or mild alcohol use disorder) or a positive drug screen test (with the exception of cannabis) verified by repeat testing
10. Lifetime history of diagnosis of schizoaffective disorder or bipolar disorder
11. Clinically significant comorbid neuropsychiatric disorders including any of the following:

    1. Current untreated or unstable major depressive disorder
    2. Clinically significant cognitive difficulties including dementia, delirium, or amnesic syndrome, within the past 2 years and would interfere with participation in the study
    3. Any other psychiatric condition that would, in the judgment of the investigator, interfere with participation in the study
12. Clinically significant or unstable medical illness/condition/disorder that would be anticipated, in the investigator's opinion, to potentially compromise patient safety or adversely affect the evaluation of efficacy, including (but not necessarily limited to) the following:

    1. Clinically significant hypotension or hypertension not stabilized by medical therapy (diastolic blood pressure > 105 mmHg)
    2. Unstable thyroid dysfunction in the past 6 months
    3. Malignant tumor within the last 5 years
    4. Neurologic conditions including the following:

    i. History of seizure disorder or condition associated with seizures ii. History of brain tumor, subdural hematoma, or other clinically significant neurological condition within the past 12 months iii. Head trauma with loss of consciousness within 12 months before screening iv. Active acute or chronic central nervous system infection v. Stroke within 6 months before screening e. Cardiac conditions including the following: i. Clinically significant cardiac arrhythmia, cardiomyopathy, or cardiac conduction defect ii. History of myocardial infarction or unstable angina within the last 3 months before screening, or clinically significant abnormality on screening or baseline electrocardiogram (ECG) including but not limited to the following: QT interval corrected for heart rate using Fridericia's formula (QTcF) > 465 msec if male or > 485 msec if female
13. Laboratory abnormality that, in the opinion of the investigator, would compromise the well-being of the patient, or any of the following laboratory abnormalities at screening or baseline:

    1. Aspartate aminotransferase or alanine aminotransferase value ≥ 2 times the upper limit of the laboratory normal reference range
    2. Hemoglobin A1c > 9%
    3. Absolute neutrophil count ≤ 1.5 × 103 μL
    4. Platelet count ≤ 75 × 103 μL
    5. Creatinine clearance < 60 mL/min
    6. Positive test result for human immunodeficiency virus, hepatitis B surface antigen, or antihepatitis C virus antibody
    7. Positive pregnancy test result
    8. Urine drug screen at screening or baseline shows a positive result for any of the tested substances (potential exceptions: results positive for benzodiazepine may not be exclusionary if the investigator confirms that such medication was medically indicated and consults the medical monitor before enrolling a patient with such a finding; results positive for Tetrahydrocannabinol (THC) may not be exclusionary in certain cases only if exclusion criterion 9 is not met and only if the medical monitor provides approval)
14. Pregnant, lactating, or breastfeeding
15. Inadequate gluteal or deltoid musculature or excessive fat, as determined by the investigator, that would interfere with IM study drug injections
16. Any contraindication for IM injections
17. Receipt of any long-acting antipsychotic medication by IM injection within 60 days before screening
18. Current involuntary hospitalization or incarceration
19. Hospitalized for more than 30 days during the 90 days before screening
20. Participation in another clinical study in which the patient received an experimental or investigational drug or agent within 6 months before screening
21. Participation in a clinical study with Risperidone ISM within 1 year before screening
22. Study site personnel and/or persons employed by the investigator or study site or is an immediate family member of such persons
23. Patients taking any prohibited concomitant medication (see Section 3.2.2.1.1) at the time of randomization visit
24. Clinically significant ocular disease or visual impairment interfering with the planned ophthalmological examinations or that in the investigator's opinion could potentially compromise patients' ocular safety
25. Patients with planned or anticipated need for ocular surgery during the treatment period of the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Litman, Principal Investigator — CBH Health LLC; Yuriy Filts, Principal Investigator — CI Lviv Regional Clinical Psychiatric Hospital. Department 25
Locations (31):
- United States (20):
  - Woodland Research Northwest, Rogers, Arkansas
  - CIMU Bellflower, Cerritos, California
  - Collaborative Neuroscience Network, LLC., Garden Grove, California
  - Synergy Research San Diego, Lemon Grove, California
  - Apostle Clinical Trials, Long Beach, California
  - NRC Research Institute, Orange, California
  - CNRI-Los Angeles LLC, Pico Rivera, California
  - CNRI-San Diego, San Diego, California
  - Galiz Research, Hialeah, Florida
  - Innovative Clinical Research Inc., Hollywood, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - CBH Health LLC, Gaithersburg, Maryland
  - Precise Research Centers MS, Flowood, Mississippi
  - Altea Research Institute, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Midwest Clinical Research Center, Dayton, Ohio
  - Carolina Clinical Triasl Inc, Charleston, South Carolina
  - Community Clinical Research Inc., Austin, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Pillar Clinical Research LLC, Richardson, Texas
- Ukraine (11):
  - Regional Clinical Hospital n.a I.I. Mechnicov, Dnipro
  - Kharkiv Regional Clinical Psychiatric Hospital, Kharkiv
  - Public Healthcare Institution "Kharkiv Regional Clinical Psychiatric Hospital No. 3", Center of Urgent Psychiatry, Kharkiv
  - Kherson Regional Psychiatric Hospital, Kherson
  - Kiev City Psychiatric Hospital No. 2, Kiev
  - Kyiv Regional Medical Association "Psykhiatriya" in Kyiv, Kiev
  - CI Lviv Regional Clinical Psychiatric Hospital. Department 20, Lviv
  - CI Lviv Regional Clinical Psychiatric Hospital. Department 25, Lviv
  - Odesa Regional Medical Centre of Mental Health, Odesa
  - Maltsev Regional Clinical Psychiatric Ho, Poltava
  - N.I. Pyrogov Vinnytsya Natl Medical University, Vinnytsia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Correll CU, Litman RE, Filts Y, Llaudo J, Naber D, Torres F, Martinez J. Efficacy and safety of once-monthly Risperidone ISM(R) in schizophrenic patients with an acute exacerbation. NPJ Schizophr. 2020 Nov 25;6(1):37. doi: 10.1038/s41537-020-00127-y. PMID 33239746

RESULTS

PARTICIPANT FLOW:
Groups:
- Risperidone in Situ Microparticle (ISM) 75 mg: Patients assigned to this arm will received 75 mg of Risperidone ISM during double-blind treatment period.
  Risperidone ISM 75 mg: Monthly IM intramuscular (IM) injection in the gluteal or deltoid muscle.
- Risperidone ISM 100 mg: Patients assigned to this arm will received 100 mg of Risperidone ISM during double-blind treatment period.
  Risperidone ISM 100 mg: Monthly IM injection in the gluteal or deltoid muscle.
- Placebo: Patients assigned to this arm will received placebo of Risperidone ISM during double-blind treatment period.
  Placebo of Risperidone ISM: Monthly IM injection in the gluteal or deltoid muscle.
Period: Overall Study
Arm/Group | Risperidone in Situ Microparticle (ISM) 75 mg | Risperidone ISM 100 mg | Placebo
Started | 144 (From 145 randomized patients in the 75 mg dose arm, one of them withdrew consent before receiving the study treatment. Due to, only 144 patients received allocated intervention.) | 146 | 147
Completed | 107 | 95 | 88
Not Completed | 37 | 51 | 59

BASELINE CHARACTERISTICS:
Population: The efficacy analysis was performed on the mITT population containing all randomized patients who received ≥1 dose of study drug with a baseline measurement and ≥1 post-baseline evaluation for the PANSS, and for whom blinding was not potentially compromised owing to a one-off error in the interactive web response system (IWRS) used for randomized treatment assignment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Risperidone ISM 75 mg | Risperidone ISM 100 mg | Placebo | Total
Number analyzed (Participants) | 129 | 129 | 132 | 390
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (10.63) | 42.6 (11.14) | 40.0 (11.35) | 41.7 (11.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 45 | 47 | 133
  Male | 88 | 84 | 85 | 257
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 10 | 19
  Not Hispanic or Latino | 123 | 126 | 122 | 371
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 58 | 63 | 59 | 180
  White | 69 | 65 | 71 | 205
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 72 | 72 | 76 | 220
  Ukraine | 57 | 57 | 56 | 170
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 27.77 (5.226) | 28.26 (5.268) | 28.19 (4.715) | 28.07 (5.065)
Years since Schizophrenia Diagnosis [Mean (Standard Deviation); unit: years] | 16.1 (10.67) | 15.7 (10.43) | 14.3 (9.74) | 15.4 (10.29)
Time since Acute Exacerbation or relapse (weeks) [Mean (Standard Deviation); unit: days] | 3 (1.95) | 3 (3.67) | 3 (1.65) | 3 (2.55)

OUTCOME MEASURES:

1. Primary Outcome: PANSS Total Score Mean Change From Baseline to Endpoint
Description: The Positive and Negative Syndrome Scale (PANSS) is a 30-item clinician-rated instrument for assessing the symptoms of schizophrenia.The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score is the sum of all 30 PANSS items and ranges from 30 to 210, with 30 indicating absence of symptoms of schizophrenia and 210 indicating extreme ratings of all 30 symptoms. Negative change from baseline scores indicate improvements in symptoms whereas higher scores mean a worse outcome.
  Endpoint is defined as study day 85 or the last post-baseline assessment if early discontinuation.
Time Frame: Day 1 (Baseline) and Day 85 (or the last post-baseline assessment)
Population: The efficacy analysis was performed on the modified Intent-to-treat (mITT) population containing all randomized patients who received ≥1 dose of study drug with a baseline measurement and ≥1 post-baseline evaluation for the PANSS, and for whom blinding was not potentially compromised owing to a one-off error in the interactive web response system (IWRS) used for randomized treatment assignment.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Risperidone ISM 75 mg | Risperidone ISM 100 mg | Placebo
Number analyzed (Participants) | 129 | 129 | 132
units on a scale | -24.6 (1.51) | -24.7 (1.54) | -11.0 (1.56)

2. Secondary Outcome: CGI-S Total Score Mean Change From Baseline to Endpoint
Description: The Clinician Global Impression - Severity (CGI-S) score is a 7-point clinician-rated scale for assessing the global severity of the illness. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Negative change from baseline scores indicate improvement in the severity of illness whereas higher scores mean a worse outcome.
  Endpoint is defined as study day 85 or the last post-baseline assessment if early discontinuation.
Time Frame: Day 1 (Baseline) and Day 85 (or the last post-baseline assessment)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Risperidone ISM 75 mg | Risperidone ISM 100 mg | Placebo
Number analyzed (Participants) | 129 | 129 | 132
units on a scale | -1.3 (0.09) | -1.3 (0.09) | -0.6 (0.09)

3. Secondary Outcome: CGI-I Score Mean at Endpoint
Description: The Clinical Global Impression - Improvement (CGI-I) Score consists of a single 7-point rating score total improvement, regardless of whether or not the change it is due entirely to drug treatment.
  Scores are: 1, Very much improved; 2, Much improved; 3, Minimally improved; 4, No change; 5, Minimally worse; 6, Much worse; or 7, Very much worse.
  Endpoint is defined as study day 85 or the last post-baseline double-blind assessment if early discontinuation.
Time Frame: Day 1 (Baseline) and Day 85 (or the last post-baseline assessment)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Risperidone ISM 75 mg | Risperidone ISM 100 mg | Placebo
Number analyzed (Participants) | 129 | 129 | 132
units on a scale | 2.5 (0.10) | 2.5 (0.10) | 3.3 (0.10)

4. Secondary Outcome: Overall Response Rate at Endpoint
Description: Overall response was defined as either PANSS total score ≥ 30% decrease from baseline, or CGI-I score of 2 (much improved) or 1 (very much improved).
  Endpoint is defined as study day 85 or the last post-baseline assessment if early discontinuation.
Time Frame: Day 85 or the last post-baseline assessment
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risperidone ISM 75 mg | Risperidone ISM 100 mg | Placebo
Number analyzed (Participants) | 129 | 129 | 132
percentage of participants | 59.7 [50.7 to 68.2] | 54.3 [45.3 to 63.1] | 20.5 [13.9 to 28.3]

5. Secondary Outcome: PANSS Response Rate at Endpoint
Description: The definition of Positive and Negative Syndrome Scale (PANSS) response was a decrease from baseline in PANSS total score of ≥ 30% (improvement of symptoms).
  Endpoint is defined as study day 85 or the last post-baseline double-blind assessment if early discontinuation.
Time Frame: Day 85 or the last post-baseline assessment
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Risperidone ISM 75 mg | Risperidone ISM 100 mg | Placebo
Number analyzed (Participants) | 129 | 129 | 132
percentage of participants | 41.9 [33.2 to 50.9] | 34.9 [26.7 to 43.8] | 9.1 [4.8 to 15.3]

6. Secondary Outcome: PANSS Positive Subscale Mean Change From Baseline to Endpoint
Description: The PANSS consisted of three subscales that contained a total of 30 symptom constructs. For each symptom construct, severity is rated on a 7-point scale, with a score of 1 indicated the absence of symptoms and a score of 7 indicated extremely severe symptoms. In positive subscale, the 7 positive symptom constructs were: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility.
  PANSS Positive Subscale Score ranges from 7 (absence of symptoms) to 49 (extremely severe symptoms).
  Endpoint is defined as study day 85 or the last post-baseline assessment if early discontinuation.
Time Frame: Day 1 (Baseline) and Day 85 (or the last post-baseline assessment)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Risperidone ISM 75 mg: Patients assigned to this arm will received Risperidone ISM 75 mg during double-blind treatment period.
  Risperidone ISM 75 mg: Monthly (once every 4 weeks) IM injection in the gluteal or deltoid muscle.
- Risperidone ISM 100 mg: Patients assigned to this arm will received Risperidone ISM 100 mg during double-blind treatment period.
  Risperidone ISM 100 mg: Monthly (once every 4 weeks) IM injection in the gluteal or deltoid muscle.
Arm/Group | Risperidone ISM 75 mg | Risperidone ISM 100 mg | Placebo
Number analyzed (Participants) | 129 | 129 | 132
units on a scale | -8.0 (0.49) | -8.7 (0.50) | -4.1 (0.50)

7. Secondary Outcome: PANSS Negative Subscale Mean Change From Baseline to Endpoint
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 indicated- absence of symptoms and a score of 7 indicated- extremely severe symptoms. The PANSS negative subscale score was the sum of the rating scores for the 7 negative scale items from the PANSS panel. The 7 negative symptom constructs were: blunted affect, emotional withdrawal, poor rapport, passive apathetic withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation and stereotyped thinking. PANSS Negative Subscale Score ranges from 7 (absence of symptoms) to 49 (extremely severe symptoms).
  Endpoint is defined as study day 85 or the last post-baseline assessment if early discontinuation.
Time Frame: Day 1 (Baseline) and Day 85 (or the last post-baseline assessment)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Risperidone ISM 75 mg | Risperidone ISM 100 mg | Placebo
Number analyzed (Participants) | 129 | 129 | 132
units on a scale | -3.8 (0.38) | -3.7 (0.39) | -1.7 (0.40)

8. Secondary Outcome: PANSS General Psychopathology Subscale Mean Change From Baseline to Endpoint
Description: The PANSS consisted of three subscales that contained a total of 30 symptom constructs. For each symptom construct, severity is rated on a 7-point scale, with a score of 1 indicated the absence of symptoms and a score of 7 indicated extremely severe symptoms. The general psychopathology scale consists of 16 items which measure somatic concern, anxiety, guilt feelings, tension, mannerisms and posturing, depression, motor retardation, uncooperativeness, unusual thought content, disorientation, poor attention, lack of judgment and insight, disturbance of volition, poor impulse control, preoccupation and active social avoidance. PANSS General Psychopathology Subscale Score ranges from 16 (absence of symptoms) to 112 (extremely severe symptoms).
  Endpoint is defined as study day 85 or the last post-baseline assessment if early discontinuation.
Time Frame: Day 1 (Baseline) and Day 85 (or the last post-baseline assessment)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Risperidone ISM 75 mg | Risperidone ISM 100 mg | Placebo
Number analyzed (Participants) | 129 | 129 | 132
units on a scale | -12.8 (0.79) | -12.4 (0.81) | -5.6 (0.82)

9. Other Pre Specified Outcome: PSP Total Score From Baseline at Each Post-baseline Assessment Time Point
Description: Personal and Social Performance Scale (PSP) total score mean change from baseline at each post-baseline assessment time point.
  The PSP is a 100-point single-item rating scale that is based on 4 domains: family and social functioning, self-care, work and socially useful activities, and disturbing and aggressive behaviors. Each domain is rated in 6 degrees of severity (absent, mild, manifest, marked, severe, very severe). On the PSP scale, higher scores indicate better social functioning: 71-100 indicates mild to no functional impairment; 31-70 varying degrees of disability and 1-30, minimal functioning needing intense support and/or supervision. Participants with a PSP total score of 71 to 100 were considered to have mild functional difficulty. Scores of 31 to 70 represented varying degrees of disability (31 to 70) and ratings of 1 to 30 indicated minimal functioning that required intense support and/or supervision.
Time Frame: Day 1 (Baseline), Days 29, 57 and 85 (or the last post-baseline assessment)
Population: The intent-to-treat (ITT) population (used for analyses of this outcome) consisted of all randomized patients who received at least 1 dose of study drug with a baseline measurement and ≥ 1 post-baseline evaluation of the PANSS. Data for both Risperidone ISM doses (75 mg and 100 mg) were pooled because this study was not powered to detect differences between doses at this endpoint and pooling this two arms the sample size increase and therefore the precision around the estimates.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Risperidone ISM: Patients assigned to this arm will received Risperidone ISM (either 75 or 100 mg) during double-blind treatment period.
  Risperidone ISM (either 75 or 100 mg): Monthly (once every 4 weeks) IM injection in the gluteal or deltoid muscle.
Arm/Group | Risperidone ISM | Placebo
Number analyzed (Participants) | 288 | 145
score on a scale
  Baseline | 49.93 [49 to 51] | 50.46 [49 to 52]
  Study Day 29 | 59.03 [58 to 60] | 55.37 [54 to 57]
  Study Day 57 | 61.33 [60 to 63] | 57.07 [55 to 59]
  Study Day 85 | 60.60 [59 to 62] | 54.54 [53 to 56]

10. Other Pre Specified Outcome: SWN-20 Total Score From Baseline at Each Post-baseline Assessment Time Point
Description: 20-item Subjective Well-Being Under Neuroleptics Treatment Scale (SWN-20) total score mean change from baseline at each post-baseline assessment time point.
  The SWN is a 38-item instrument to measure subjective effects of neuroleptic medications in patients with schizophrenia and consists of 20 positive statements and 18 negative statements. The short form of the SWN, the 20-item SWN-20, was developed in order to allow for quick assessment of subjective side effects in a clinical setting. Like in the original SWN, with the SWN-20 the patient is asked to rate well-being items that have been identified as related to antipsychotic treatment on a 6-point scale ranging from "Not at all" to "Very much." The SWN-20 is scored on a scale ranging from 20 to 120, with higher scores indicating better health-related quality of life (HRQL). The SWN-20 contains five 4-item subscales: mental functioning, self-control, emotional regulation, physical functioning, and social integration. Eac
Time Frame: Day 1 (Baseline), Days 29, 57 and 85 or the last post-baseline assessment
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Risperidone ISM | Placebo
Number analyzed (Participants) | 288 | 145
score on a scale
  Baseline | 80.86 [79 to 83] | 80.28 [78 to 83]
  Day 29 | 86.90 [85 to 89] | 83.23 [81 to 86]
  Day 57 | 88.26 [87 to 90] | 86.32 [83 to 89]
  Day 85 | 89.14 [88 to 91] | 85.50 [83 to 88]

11. Other Pre Specified Outcome: Plasma PK Parameters
Description: Plasma PK Parameters of Risperidone Active Moiety
  Cmax values are estimated and based on the plasma level of Day 3 for each dosing Interval; Cmin are the trough levels of Day 29, which is at the end of each dosing Interval;
Time Frame: Day 3 and Day 29 after Dose 1, 2 and 3
Population: Pharmacokinetic (PK) population included patients in the safety population who have at least 1 measurement plasma concentration value.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Risperidone ISM 75 mg: Risperidone ISM 75 mg dose
- Risperidone ISM 100 mg: Risperidone ISM 100 mg dose
Arm/Group | Risperidone ISM 75 mg | Risperidone ISM 100 mg
Number analyzed (Participants) | 144 | 146
ng/mL
  Dose 1/Estimated Cmax/Day 3 | 27.61 (19.992) | 32.00 (16.802)
  Dose 1/Estimated Cmin/Day 29 | 19.21 (13.076) | 26.71 (14.960)
  Dose 2/Estimated Cmax/Day 3 | 38.95 (22.381) | 53.44 (23.840)
  Dose 2/Estimated Cmin/Day 29 | 17.46 (13.418) | 27.23 (14.070)
  Dose 3/Estimated Cmax/Day 3 | 37.16 (19.504) | 50.09 (22.242)
  Dose 3/Estimated Cmin/Day 29 | 20.16 (16.847) | 26.14 (16.343)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected in all visits of the study, from the patient's signature of informed consent form through the end of study for each subject: Screening visit, Baseline (Day 1), Day 3, 4, 8, 15, 22, 29, 31, 43, 57, 59, 71, 85 and follow-up visit (Day 99).
Description: The analysis was performed in the Safety Population, which includes all patients who received at least 1 dose of the study drug. 437 patients were included in the safety population.
Arm/Group | Risperidone ISM 75 mg | Risperidone ISM 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/144 | 0/146 | 0/147
Serious Adverse Events (participants affected / at risk) | 2/144 | 5/146 | 5/147
Other Adverse Events (participants affected / at risk) | 101/144 | 119/146 | 48/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risperidone ISM 75 mg (N=144) | Risperidone ISM 100 mg (N=146) | Placebo (N=147)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 1 (1) | 2 (2) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risperidone ISM 75 mg (N=144) | Risperidone ISM 100 mg (N=146) | Placebo (N=147)
Tachycardia (Cardiac disorders) | 2 (2) | 4 (4) | 0 (0)
Hyperprolactinaemia (Endocrine disorders) | 8 (8) | 13 (13) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2)
Injection site pain (General disorders) | 8 (10) | 4 (5) | 5 (7)
Nasopharyngitis (Infections and infestations) | 5 (5) | 4 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 7 (7) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 4 (4) | 3 (3)
Blood prolactin increased (Investigations) | 13 (15) | 21 (22) | 0 (0)
Blood triglycerides increased (Investigations) | 4 (4) | 3 (3) | 1 (2)
Weight increased (Investigations) | 10 (10) | 8 (8) | 3 (3)
Akathisia (Nervous system disorders) | 6 (6) | 11 (13) | 3 (3)
Dizziness (Nervous system disorders) | 5 (5) | 6 (6) | 4 (4)
Dystonia (Nervous system disorders) | 4 (4) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 15 (17) | 12 (12) | 5 (6)
Somnolence (Nervous system disorders) | 4 (5) | 8 (8) | 4 (4)
Insomnia (Psychiatric disorders) | 4 (4) | 6 (8) | 6 (8)
Schizophrenia (Psychiatric disorders) | 3 (3) | 3 (4) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor does not object to publication by the Institution of the results of the Trial based on information collected/generated by the Institution. The Institution will provide Sponsor an opportunity to review any proposed publication before it is submitted. If the Trial is part of a multi-center trial, the Institution agress that the first publication is to be a joint publication involving all Trials sites.

DOCUMENTS (3):
  • Study Protocol (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT03160521/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT03160521/SAP_001.pdf
  • Informed Consent Form (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT03160521/ICF_003.pdf